CLINICAL TRIAL: NCT05611554
Title: Parental Stress, Health and Disabilities. A Training Programme in Psychological Flexibility During COVID 19
Brief Title: Effects of an ACT-based Psychological Treatment in Relatives of People With Intellectual Disabilities
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIPI/21/091
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Parent-Child Relations; Parental Stress
Keywords: stress; acceptance and commitment therapy; health; parent-child relations

STUDY DESIGN:
Intervention Model Description: Randomization assigned participants to 2 arms:
  1. Treatment
  2. Waiting list
Masking Description: The participants were aware of the existence of the two conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Psychological intervention will consist in an 3-session group ACT-based treatment.
  Interventions: Behavioral: ACT
- Waiting List (No Intervention): Participants assigned to Waiting List arm waited for 5 months before receiving treatment (i.e., after completing the measures they continued in the study and received Psychological intervention five months later)

INTERVENTIONS:
Behavioral: ACT — Psychological intervention focused on (a) values clarification, (b) defusion strategies, (c) training in flexible attention to the present moment (mindfulness), and (d) committed action and psychological acceptance through metaphors and experiential exercises.
  Arms: Treatment

SUMMARY:
Investigation of the efficacy of Acceptance and Commitment Therapy (ACT) for the psychological treatment of parental stress in relatives of people with intellectual disabilities

DETAILED DESCRIPTION:
After being informed about the study, all patients giving written informed consent will be assessed to determine eligibility for study entry.

Patients who meet eligibility requirements will receive psychological intervention consisting in 3-session group ACT-based treatment.

The participants will be assessed through self-report instruments before and after treatment and at 3 months follow-up.

The clinical trial will include a control group.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* High level of understanding of Spanish
* Having children diagnosed with intellectual disability

Exclusion Criteria:

* Current psychological and/or psychiatric treatment,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2023-02-15 (Estimated)

PRIMARY OUTCOMES:
Change in Perceived Stress Scale (PSS) | Change from Baseline perceived stress at 4 months
  Perceived Stress Scale (PSS) is a one-dimensional scale with 14 items that are answered on a Likert-type scale ranging from 0 (Never) to 5 (Very often). The direct scores range from 0 to 56; higher scores indicate higher perceived stress and worse outcome.

SECONDARY OUTCOMES:
Change in Parental Acceptance Questionnaire (6-PAQ) | Change from Baseline Psychological Inflexibility at 4 months
  Parental Acceptance Questionnaire (6-PAQ) is a 16-item questionnaire on a Likert-type scale with four answer options in a range from 1 (Strongly Disagree) to 4 (Strongly Agree) that assesses six processes related to psychological flexibility (being present, values, committed action, self as context, cognitive defusion, and acceptance) and three flexible response styles (opened, centred and committed). The scores vary from 16 to 64; the higher the score, the higher psychological inflexibility levels and worse outcome.
Change in Psychological Health Questionnaire (GHQ-12) | Change from Baseline Psychological Well-Being at 4 months
  Psychological Health Questionnaire (GHQ-12) contains 12 items on a Likert-type scale with four answer options in a range from 0 (Strongly Disagree) to 3 (Strongly Agree). Higher scores indicate lower levels of psychological well-being and worse outcome.
Change in White Bear Suppression Inventory (WBSI) | Change from Baseline thoughts suppression at 4 months
  White Bear Suppression Inventory (WBSI) evaluates the tendency to suppress unwanted thoughts. It is a Likert scale of 15 items with five response options ranging from 1 (Completely Disagree) to 5 (Completely Agree). Scores range from 15 to 75. Higher scores indicate a stronger thought suppression tendency and worse outcomes.
Change in Behavioural self-monitoring | Change from Baseline punitive-hostile and supportive-companion behaviours at 1 month.
  Behavioral self-monitoring captures behaviour change. Family members recorded a daily estimation of the frequency of two categories of behaviours: punitive-hostile behaviours from family members to children with disabilities (e.g., shouting, punishments, insults, or aggressions) and supportive-companion behaviours (e.g., helping, shared leisure and recognition or compliments). A Likert-type scale was used to estimate frequency, with values from 0 to 4 (0= never; 1= almost never; 2= sometimes; 3= often; and 4= always) Participants completed daily self-monitoring, starting one week before the intervention (forming the baseline scenario) until one week after the intervention, obtaining a total of 4 measures. Higher scores in punitive-hostile behaviours indicate higher levels of punitive-hostile behaviours and worse outcome. Higher scores in supportive-companion behaviours indicate higher levels of supportive-companion behaviours and better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Montesinos, PhD, Principal Investigator — Universidad Europea de Madrid
Locations (1):
- Universidad Europea de Madrid, Madrid, Villaviciosa de Odón, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT05611554/Prot_000.pdf
  • Informed Consent Form (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT05611554/ICF_001.pdf